CLINICAL TRIAL: NCT04761731
Title: A Single Center, Single Arm, Open-label Study to Evaluate the Efficacy and Safety of Tacrolimus Modified Release, ADVAGRAF® After Treatment With a Tacrolimus in New Liver Transplant Recipients
Brief Title: To Evaluate the Efficacy and Safety of ADVAGRAF® After Treatment With a Tacrolimus in New Liver Transplant Recipients
Acronym: Assign
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Linical Korea (Industry)
Collaborators: Astellas Pharma Korea, Inc. (Industry); National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Assign
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Liver Transplantation
Keywords: ADVAGRAF®; liver transplantation; tacrolimus
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADVAGRAF® (Experimental): One arm: Treatment conversion will take place from twice daily tacrolimus to once daily tacrolimus (ADVAGRAF) 3 months after transplant in new liver transplant recipients.
  Interventions: Drug: ADVAGRAF®

INTERVENTIONS:
Drug: ADVAGRAF® — Administration method The total daily dose of tacrolimus will be converted to 1:1 (mg:mg) and the total daily dose of ADVAGRAF® will be administered only once daily in the morning, starting from Day 1 (at least one hour before breakfast or 2 to 3 hours after breakfast).
  * Dose adjustment after conversion On Day 1, the total dose will be converted to 1:1. It is recommended to check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~8ng/ml for 0 to 3 months and then at 5ng/ml or below for 3 to 6 months of study treatment.
  * Duration of treatment The investigational product will be administered for 24 weeks.
  Other Names: tacrolimus

SUMMARY:
This study's objective is to evaluate the incidence rate of acute rejection reactions after 24 weeks treatment with ADVAGRAF® following 3 months treatment with tacrolimus in new liver transplant recipients.

Treatment conversion will take place from twice daily tacrolimus to once daily tacrolimus (ADVAGRAF) 3 months after transplant in new liver transplant recipients.

DETAILED DESCRIPTION:
This is single center,open-label study with ADVAGRAF® Primary endpoint is Incidence rate of biopsy confirmed acute rejection reactions within 24 weeks following conversion+ Incidence rate of acute rejection reactions (%) = number of subjects with at least one acute rejection reaction 1)/total number of subjects in the relevant analysis set * 100 Only those acute rejection reactions confirmed by biopsy will be acceptable as acute rejection reactions.

Administration method is following The total daily dose of tacrolimus will be converted to 1:1 (mg:mg) and the total daily dose of ADVAGRAF® will be administered only once daily in the morning, starting from Day 1 (at least one hour before breakfast or 2 to 3 hours after breakfast).

* Dose adjustment after conversion On Day 1, the total dose will be converted to 1:1. It is recommended to check the blood concentration of tacrolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 5~8ng/ml for 0 to 3 months and then at 5ng/ml or below for 3 to 6 months of study treatment.
* Duration of treatment The investigational product will be administered for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* When the Subjects agree informed consent form, Subject should be More than 20 years of age

  * Those who are transplanated liver at a minimum of 10 weeks or Maximum of 14 weeks of baseline

    * Average of tacrorimus trough level is 3-10 ng/mL from transplanted date to before baseline.

      * Female subjects of child bearing potential must have a negative urine or serum pregnancy test prior to enrolment and at the end of study and must agree to practice effective birth control during the study.(The oral contraceptive pill is not allowed to take a female subject) ⑤Subjects are stable clinically in the opinion of the investigator. ⑥Subjects capable of understanding the purpose and risks of the study, having been fully informed and has given written informed consent to participate in the study

Exclusion Criteria:

* Subjects having previously received an organ transplant excluding liver transplant. Or Subjects receiving an auxiliary graft or in whom a bio-artificial liver(cell system) has been used.

  * Acute rejection from transplanted date to before baseline

    * Subjects diagnosed new malignant tumor after liver transplantation, with the exception of basalioma or squamous cell carcinoma of the skin that has been treated successfully.

      * Subjects allergic to tacrolimus or investigational product.

        * Subjects are unstable clinically state in the opinion of the investigator.

          * Subjects with any form of substance abuse, psychiatric disorder or condition which, in the opinion of the investigator, may complicate communication with the investigator.

            ⑦Subjects participating or having participated in another clinical trial and/or those taking or having taken an investigational / non-registered drug in the past 28 days.

            ⑧Subjects taking forbidden concomitant medications or within 28 days prior to enroll.
            * Subjects who are pregnant or breast-feeding mother.

              ⑩Subjects known to be HIV positive.

              ⑪Subjects unlikely to comply with the visits scheduled in the protocol.

              ⑫Subjects with renal dysfunction on the investigator's point of view or serum creatinine > 1.6mg/dL or GFR(MDRD)<30mL/min in the baseline.

              ⑬Hepatic dysfunction: rising more than triple the normal range of SGPT/ALT and/or SGOT/AST and/or bilirubin, hepatic cirrhosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence rate of biopsy confirmed acute rejection | 24 weeks within
  Incidence rate of acute rejection reactions (%) = number of subjects with at least one acute rejection reaction 1)/total number of subjects in the relevant analysis set * 100

SECONDARY OUTCOMES:
Severity of biopsy confirmed acute rejection | within 24 weeks
  Severity of acute rejection reactions is defined as the highest severity in a subject who had at least one acute rejection reaction.
Survival rates of subjects and transplanted organs | at 24 weeks
  The survival rate of transplant organs is determined by the loss of transplant organs in the 24th week. Transplant organ loss is defined as re-transplant surgery or death. The date of the transplant's disappearance is the first time one of these events has occurred.
compliance | at 24 weeks
  The dosage compliance level is checked by the questionnaire at each visit based on the total amount of the IPs that should have been taken.

CONTACTS AND LOCATIONS:
Overall Officials: seoung hoon Kim, doctoral, Principal Investigator — National Cancer Center, Korea